CLINICAL TRIAL: NCT02023853
Title: The Use of Erythritol Powder and Locally Derived Metronidazole for the Non-surgical Treatment of Peri-implant Mucositis and Peri-implantitis.
Brief Title: Non Surgical Treatment of Periimplantitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Proed, Torino, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Proed.08.2013.periimplantitis
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis
MeSH Terms: conditions — Peri-Implantitis | interventions — High-Energy Shock Waves; Erythritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasonic, erythritol, metronidazole gel (Experimental)
  Interventions: Procedure: ultrasonic; Procedure: erythritol; Drug: metronidazole gel

INTERVENTIONS:
Procedure: ultrasonic
Procedure: erythritol
Drug: metronidazole gel

SUMMARY:
20 consecutive adult implant patients, presenting the signs of peri-implant mucositis (probing depth ≥4 mm combined with bleeding and/or pus on probing) or initial peri-implantitis (probing depth ≥4 mm, bleeding and suppuration plus radiographic loss of supporting bone ≤30% compared with the situation after implant placement) will be included.

Sites will be treated by ultrasonic debridement of the pocket, performed using a piezoceramic ultrasonic device. For the purpose, a Tip will be connected to the Handpiece Led (5 minutes/pocket) . Then, it will be followed by the subgingival use of erythritol powder applied by the use of Handpiece connected to an airflow unit 2x5 seconds/pocket. At this time the subgingival delivery of metronidazole gel will be provided. After instrumentation, patients will rinse with chlorhexidine 0.20% 3 times/day for 2 weeks.

At baseline, 1 month, 3 months and 6 months the following parameters will be evaluated: Probing Pocket depth (PPD), Bleeding on Probing (BoP), Clinical Attachment Level (CAL).

ELIGIBILITY:
Inclusion Criteria:

* adult patients suffering from peri-implant mucositis or peri-implantitis

Exclusion Criteria:

* Heavy smokers current pregnant history of malignancy long-term steroidal or antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
probing pocket depth change | baseline, 6 months
bleeding on probing change | baseline, 6 months
clinical attachment level change | baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Cardaropoli, DDS, Principal Investigator — Proed, Torino, Italy
Locations (1):
- PROED, Institute for Professional Education in Dentistry, Torino, Italy